CLINICAL TRIAL: NCT06434662
Title: A Phase II Study of the Safety and Efficacy of Mitoxantrone Hydrochloride Liposome Injection, Cytarabine and Venetoclax in Patients With Relapsed/Refractory AML
Brief Title: Mitoxantrone Hydrochloride Liposome Injection, Cytarabine Combined With Venetoclax in the Treatment of R/R AML
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: CSPC Zhongnuo Pharmaceutical (Shijiazhuang) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DED-AML-K13
Record Dates: First submitted 2024-05-10; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-03

CONDITIONS: Relapsed/Refractory Acute Myeloid Leukaemia; Myeloid Malignancy
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MAV regimen (Experimental): mitoxantrone hydrochloride liposome injection, cytarabine combined with venetoclax
  Interventions: Drug: mitoxantrone hydrochloride liposome; Drug: Cytarabine; Drug: Venetoclax

INTERVENTIONS:
Drug: mitoxantrone hydrochloride liposome — Mitoxantrone hydrochloride liposome (24 mg/m^2) on day 1, every 4 weeks
Drug: Cytarabine — Cytarabine (1.0 g/m^2, q12h ) on day 1,3,5, every 4 weeks
Drug: Venetoclax — Venetoclax 100 mg on day 2，200 mg on day 3，400 mg on day 4-10, every 4 weeks

SUMMARY:
The goal of this study is to evaluate the efficacy and safety of a combination regimen of mitoxantrone hydrochloride liposome injection, cytarabine and venetoclax (MAV) in the treatment of relapsed or refractory (R/R) AML. It will also tentatively explore the correlation between different biological characteristics and therapeutic efficacy. The main questions it aims to answer are:Dose the combination regimen of MAV enhanced the composite complete remission in R/R AML? Participants will receive laboratory tests of bone marrow and blood specimens at regular times after MAV treatment.

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) is a highly aggressive hematologic malignancy with a poor prognosis. The "3+7" regimen, combining anthracyclines with cytarabine, remains the standard treatment for first line treatment. However, about 20% of patients will develop into primary refractory disease, and more than 50% of patients who achieved complete remission will eventually relapse. For patients with R/R AML, there is currently no established standard treatment. Combining the third drugs with "3+7" regimen is one of the clinical exploration directions.

The purpose of this prospective, single-center, single-arm, pahse II study is to evaluate the efficacy and safety of a combination regimen of mitoxantrone hydrochloride liposome injection, cytarabine and venetoclax in the treatment of R/R AML. All participants will receive MAV treatment including 24 mg/m2 mitoxantrone hydrochloride liposome on day 1, 1.0 g/m2 q12h cytarabine on day 1,3,5 and 400 mg venetoclax on day 2-10 with a dose escalation on day 2-4. Each cycle consists of 4 weeks. A maximum of 2 cycles of therapy are planned.

ELIGIBILITY:
Inclusion Criteria:

1. Each subject must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and are willing to participate in the study.
2. Age ≥18.
3. Clinically diagnosed relapsed/refractory AML, excluding acute promyelocytic leukemia.

   1. Initial treatment patients who failed after 2 courses of treatment with standard regimen.
   2. Bone marrow blasts≥5% after the first CR/CRi, or reappearance of blasts in the blood in at least 2 peripheral blood samples at least one week apart, or leukemia cell infiltration appeared in extramedullary without treatment.
   3. First conversion from MRD negativity to MRD positivity without treatment.
4. Physical status score of Eastern Oncology Collaboration Group (ECOG) : 0-2.
5. Researchers determined that the patients could tolerate intensive chemotherapy.
6. Life expectancy > 3 months.
7. AST/ALT≤2.5 ULN (for subjects with hepatic infiltration≤5 ULN); Total bilirubin≤1.5 ULN (for subjects with hepatic infiltration≤3 ULN); Serum creatinine≤1.5 ULN.

Exclusion Criteria:

1. Previous anti-tumor therapy meets one of the following criteria:

   1. Prior therapy with mitoxantrone or mitoxantrone liposome;
   2. Prior therapy with doxorubicin or anthracyclines, and the cumulative dose of doxorubicin > 360 mg/m^2 (1 mg doxorubicin was equivalent to 2 mg daunorubicin or 0.5 mg idarubicin);
   3. Have received other anti-tumor therapy (including chemotherapy, targeted therapy, hormone therapy, Chinese medicines with anti-tumor activity, except those that do not affect the efficacy of the study as determined by the investigator) or participated in other clinical trials and received clinical trial drugs within 4 weeks or 5 half-lives of the drug before the study;
2. Cardiovascular diseases, including but not limited to:

   1. QTc interval >480 ms or long QTc syndrome in screening;
   2. Complete left bundle branch block, 2 or 3 grade atrioventricular block;
   3. Requiring treatment of serious and uncontrolled arrhythmia;
   4. New York Heart Association（NYHA≥3;
   5. Cardiac ejection fraction (EF) was less than 50%;
   6. Myocardial infarction, unstable angina pectoris, severe unstable ventricular arrhythmia or any other history of arrhythmia or clinically serious pericardial disease that requires treatment within the first 6 months of enrollment, or electrocardiographic evidence of acute ischemic or active conduction system abnormalities.
3. Central nervous system leukemia;
4. Previous or current occurrence of other malignancies (in addition to non-melanoma basal cell carcinoma of the skin that is effectively controlled, breast/cervical carcinoma in situ, and other malignancies that have been effectively controlled without treatment within the past five years).
5. Subjects are suffering from any other uncontrollable disease (including but not limited to: uncontrolled diabetes and hypertension, and advanced infection);
6. HIV infection.
7. HBsAg or HBcAb positive, with HBV-DNA≥1x10^3 copies/mL; or HCV-RNA≥1x10^3 copies/mL;
8. A history of immediate or delayed allergy to similar drug and excipients of the investigate drug.
9. Pregnant, lactating female or subjects who refuse to use effective contraception during the study.
10. With a history of severe neurological or psychiatric illness.
11. Not suitable for this study as decided by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Composite complete remission (CRc) rate | At the end of each cycle (each cycle is 28 days), up to 2 cycles
  Blast rate lower than 5% with or without peripheral blood cell recover

SECONDARY OUTCOMES:
Overall response rate (ORR) | At the end of each cycle (each cycle is 28 days), up to 2 cycles
  Response is assessed according to the the European LeukemiaNet (ELN) 2022 criteria
Relapsed free survival (RFS) | up to 12 months
  Defined only for patients achieving CR or CRi; measured from the date of achievement of remission until the date of hematologic relapse or death from any cause;
Event free survival (EFS) | up to 12 months
  Defined for all patients in a trial; measured from day 1 of treatment to the date of treatment failure, hematologic relapse from CR/CRi or death from any cause, whichever occurs first;
overall survival (OS) | up to 12 months
  Defined for all patients in a trial; measured from day 1 of treatment to the date of death from any cause;
Rate of CR without minimal residual disease (CR MRD-) | At the end of each cycle (each cycle is 28 days), up to 2 cycles
  Percentage of participants who achieve a CR MRD- as defined by investigators based on ELN 2022 criteria; MRD level is detected by flow cytometry which value <0.1% is defined as negtive;
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From day 1 of treatment to 28 days after the last dose
  The safety of the drug was evaluated by NCI-CTC AE 5.0 standard.Hematologic and non-hematologic toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Jin, M.D., Principal Investigator — Zhejiang University
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No